CLINICAL TRIAL: NCT07054528
Title: Multicentre Real-life Data Collection Study With CareMin650™ in the Prevention and Treatment of Oral Mucositis and Radio- and/or Chemo-induced Dermatitis
Acronym: NéoPBM
Status: Active, not recruiting | Type: Observational
Sponsor: Centre Hospitalier de Valenciennes (Network)
Responsible Party: Sponsor
Other Study IDs: 2024-03-01
Record Dates: First submitted 2025-06-02; First posted 2025-07-08 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Oral Mucositis (Ulcerative); Oral Mucositis (Ulcerative) Due to Antineoplastic Therapy; Oral Mucositis (Ulcerative) Due to Radiation; Dermatitis
Keywords: Oncology; Photobiomodulation; oral mucositis; dermatitis; chemotherapy; radiotherapy
MeSH Terms: conditions — Stomatitis; Ulcer; Dermatitis; Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Most patients with cancer or haematological malignancies who receive chemotherapy - broadly defined to include targeted therapies and immunotherapy - and/or external beam radiotherapy may experience serious and disabling adverse events related to these treatments.

Mucositis and radiodermatitis are a frequent and disabling complication of cancer and haematological malignancy treatments: chemotherapy (in the broadest sense: includes immunotherapy, targeted therapies) and/or radiotherapy, having a considerable impact on patients' quality of life.

Mucositis is linked to lesions that occur in epithelial and connective tissues in response to a complex cascade of biological events involving the cellular elements of the mucosa.

All these consequences make for an inadequate care pathway (hospitalisations and urgent care, complications, decompensations of comorbidities) and considerably increase the financial cost of patient care. Management strategies are perfectly codified, and photobiomodulation is now recommended internationally with a high level of evidence for the prevention and treatment of oral mucositis and radiodermatitis.

Photobiomodulation (PBM), previously known as low-level laser therapy, has been used for decades in numerous therapeutic indications, based on major scientific knowledge and significant scientific and technological developments Including in fields such as aerospace or military medicine.

CareMin650™ is a photobiomodulation medical device marketed since 2020 and indicated for the treatment of oral mucositis and radiodermatitis.

The aim of the registry is to describe the real-life use of CareMin650™ in France in the preventive and curative treatment of radio and/or chemo-induced oral mucositis and radiodermatitis.

ELIGIBILITY:
Inclusion Criteria:

* Any adult patient over 18 years of age
* Patient treated with the CareMin650™ photobiomodulation device, as a preventive or curative measure for oral mucositis and/or radiodermatitis induced by chemotherapy (in the broadest sense: includes targeted therapies, immunotherapy) and/or radiotherapy, as part of their routine management for any type of cancer or haematological malignancy, whatever the stage and prognosis of the disease
* Information note sent to the patient and record of the patient's or legal representative's (guardian's) non-objection
* Membership of a social security scheme

Exclusion Criteria:

* Pregnant women
* Patient with severe cognitive impairment rendering him/her incapable of expressing non-objection to participation in the study.
* If the patient is under guardianship or curatorship: objection from the guardian/curator.
* Patient with a known allergy to polyurethane
* Patient taking part in a clinical study involving medicinal or non-medicinal therapies to treat or prevent oral mucositis or radiodermatitis.
* Patients physically unable to apply Ora-Pad and Derma-Pad devices (e.g. limited mouth opening).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Most patients with cancer or haematological malignancies receiving chemotherapy and presenting with oral mucositis and/or radio- and/or chemo-induced dermatitis will have some form of oral mucositis.
Sampling Method: Probability Sample
Enrollment: 33000 (Estimated)
Dates: Start 2025-06-20 (Actual); Primary Completion 2034-10-30 (Estimated); Study Completion 2034-10-30 (Estimated)

PRIMARY OUTCOMES:
Evaluation of the evolution of the severity of radio- and/or chemo-induced oral mucositis lesions and radiodermatitis during preventive or curative treatment with CareMin650™ between the first and last session. | Measured at the first of photobiomodulation and at the last session (Week 12)
  * Grading of lesions according to WHO scales for oral mucositis
    0 - No lesion
    1 - Erythema - moderate pain 2 - Moderate ulceration - solid food 3- Severe ulceration - liquid food 4 - Severe ulceration - no oral feeding
  * Grading of lesions according to WHO scales for radiodermatitis
    0 - No lesion
    1. - Mild erythema or dry desquamation
    2. - Moderate to vivid erythema - localized moist desquamation in folds - moderate edema
    3. - Localized moist desquamation other than in folds - minor bleeding due to light trauma or abrasion
    4. - Ulceration or necrosis - spontaneous bleeding - indication for grafting

SECONDARY OUTCOMES:
Assessment of the satisfaction of professionals using the CareMin650™ | At last photobiomodulation session Week 12
  Assessment of the satisfaction of CareMin650™ users (nurses, doctors, radio manipulators) :
  1. Ease of device installation (4-point Likert scale)
     * Very satisfactory
     * Somewhat satisfactory
     * Rather unsatisfactory
     * Not at all satisfactory
  2. Conditions for programming the device (4-point Likert scale) How did the installation of the device go?" "Very easy"; "Rather easy", "Rather difficult"; "Very difficult".
  3. Overall assessment of device ergonomics (ease of use) (4-point Likert scale) In your opinion, using the device is " " Very convenient " ; " Rather convenient " ; " Rather inconvenient " ; " Not at all convenient "
Assessment of patient satisfaction | At last photobiomodulation session week12
  Assessment of patient satisfaction following CareMin650™ sessions:
  * Level of constraint related to PBM (4-level Likert scale)
  * Existence of pain when applying the device (4-point Likert scale)
  * Discomfort during sessions (4-point Likert scale)
  * Overall satisfaction with duration of sessions
Description of the conditions of real-life use of CareMin650™ | At last session of photobiomodulation week 12
  Description of the conditions of real-life use of CareMin650™ :
  * Therapeutic objective
  * Nature of carer carrying out PBM treatment
  * Average number of sessions performed per week
  * Total number of sessions performed
  * Administration before, during or after chemotherapy and/or radiotherapy
  * Dose prescribed according to therapeutic objective (preventive/curative)
  * Used alone or in combination with another PBM device
Assessment of the clinical benefit of CareMin650™ in the management of oral mucositis for the patient | At last session of photobiomodulation week 12
  Assessment of the clinical benefit of CareMin650™ in the management of oral mucositis for the patient / QUESTIONNAIRES ABOUT :
  * Ability to feed: solid and liquid oral nutrition, liquid/semi-liquid oral nutrition, enteral tube feeding
  * Medicinal treatments for oral mucositis (type of treatment, dosage, duration)
  * Related medicinal treatments, in particular analgesics and psychotropic drugs (nature of treatments, names of molecules, dosages, duration of treatment, and possible modifications during photobiomodulation treatment)
  * Evaluation of oral pain by Visual Analogue Scale before and after each session
  * Duration of each session

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier de Valenciennes, Valenciennes, France, France